CLINICAL TRIAL: NCT00932061
Title: Developing Biomarkers for Fibromyalgia
Acronym: Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: The Dana Foundation (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Richard Harris, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Hum 00010061; F017513; Sponsor(DOD) W81XWH-07-20050
Record Dates: First submitted 2009-06-25; First posted 2009-07-02 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Healthy controls; Acupuncture; Sham Acupuncture; fMRI; Biological marker
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional Acupuncture (Active Comparator): Acupuncture sites will be used for active intervention.
  Interventions: Other: Traditional Acupuncture
- Sham Treatment (Sham Comparator): Sham acupuncture is used.
  Interventions: Other: Sham Treatment

INTERVENTIONS:
Other: Traditional Acupuncture — Fibromyalgia subjects will be randomized to receive 9 acupuncture treatments over the course of four weeks.
  Subjects enrolled in the study may have 1) only fMRI or 2) fMRI scans and PET scans, depending on their eligibility criteria.
  Arms: Traditional Acupuncture
Other: Sham Treatment — Fibromyalgia subjects will be randomized to receive 9 sham treatments over the course of four weeks.
  Subjects enrolled in the study may have 1) only fMRI or 2) fMRI scans and PET scans, depending on their eligibility criteria.
  Arms: Sham Treatment

SUMMARY:
The hypothesis of this study is that biological markers are present in the body that are good indicators of chronic pain. Eligible participants will be assessed at baseline and after receiving a series of acupuncture or "sham" acupuncture (something that resembles, but is not, active acupuncture) sessions. If the subject qualifies for the investigators' research and are subsequently enrolled in this study, they will be randomly assigned (like the flip of a coin) to one of these two groups. Acupuncture, as previously shown by this group, leads to improvements in both clinical and evoked pain associated with fibromyalgia. The study involves two magnetic resonance imaging (MRI) brain scans, one at the beginning and one at the end of the study. Another optional portion of the study would involve 2 PET (positron emission tomography) scans of the subject's brain, one at the beginning and one at the end of the study; this type of scan allows us to get more specific information about the subject's brain function during an acupuncture session.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Fibromyalgia Volunteers:

* Has met American College of Rheumatology (1990) criteria for the diagnosis of fibromyalgia for at least 1 year
* Chronic pain more than 50% of days
* Willing to limit introduction of any new medications or treatments for fibromyalgia during the study
* Able to attend study visits up to three times weekly
* Right-handed
* Be capable of giving written informed consent

Inclusion Criteria for Healthy Volunteers:

* Willing to refrain from alcohol intake for 48 hours prior to brain scans
* Be right handed
* Be capable of giving written informed consent

PET Inclusion Criteria:

* Willing to refrain from alcohol intake 48 hours prior to brain scans
* Capable of giving written consent

Exclusion Criteria:

Exclusion Criteria for Fibromyalgia Volunteers:

* Knowledge that could prevent "blinding" of the participant to the study interventions (including previous acupuncture treatment)
* Presence of a known coagulation abnormality, thrombocytopenia, or bleeding diathesis that may preclude the safe use of acupuncture
* Autoimmune or inflammatory disease (in addition to fibromyalgia) that causes pain (e.g., rheumatoid arthritis, systemic lupus erythematosus, inflammatory bowel disease)
* Daily use of narcotic pain-relievers
* History of substance abuse
* Simultaneous participation in other therapeutic trials
* Pregnant or breastfeeding
* Current severe psychiatric illness (e.g., schizophrenia, major depression with suicidal ideation)
* Condition that may make exposure to fMRI medically inadvisable
* Any condition that may prevent satisfactory completion of the study protocol

Exclusion for Healthy Volunteers:

* Autoimmune or inflammatory disease (in addition to fibromyalgia) that causes pain (e.g., rheumatoid arthritis, systemic lupus erythematosus, inflammatory bowel disease)
* Having met the ACR criteria for FM
* Simultaneous participation in other therapeutic trials
* Pregnant or breastfeeding
* Current severe psychiatric illness (e.g., schizophrenia, major depression with suicidal ideation)
* Condition that may make exposure to fMRI medically inadvisable
* Any condition that may prevent satisfactory completion of the study protocol

PET Exclusion Criteria:

* Meets any of the fMRI exclusion criteria
* Current major depression
* Condition that may make exposure to PET medically inadvisable

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2008-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
fMRI signal | pre treatment - week 1
PET signal | pre treatment - week 1
H-MRS Glutamate | pre treatment - week 1
fMRI signal | post treatment - week 5
PET signal | post treatment - week 5
H-MRS - Glutamate | post treatment - week 5

SECONDARY OUTCOMES:
Pain | pre treatment - week 1
Pain | post treatment - week 5

CONTACTS AND LOCATIONS:
Overall Officials: Richard Harris, Ph.D., Principal Investigator — Univeristy of Michigan, Chronic Pain & Fatigue Research Center
Locations (1):
- University of Michigan, Chronic Pain and Fatigue Research Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Harris RE, Zubieta JK, Scott DJ, Napadow V, Gracely RH, Clauw DJ. Traditional Chinese acupuncture and placebo (sham) acupuncture are differentiated by their effects on mu-opioid receptors (MORs). Neuroimage. 2009 Sep;47(3):1077-85. doi: 10.1016/j.neuroimage.2009.05.083. Epub 2009 Jun 6. PMID 19501658
- [Result] Harris RE, Sundgren PC, Pang Y, Hsu M, Petrou M, Kim SH, McLean SA, Gracely RH, Clauw DJ. Dynamic levels of glutamate within the insula are associated with improvements in multiple pain domains in fibromyalgia. Arthritis Rheum. 2008 Mar;58(3):903-7. doi: 10.1002/art.23223. PMID 18311814
- [Result] Harris RE, Clauw DJ, Scott DJ, McLean SA, Gracely RH, Zubieta JK. Decreased central mu-opioid receptor availability in fibromyalgia. J Neurosci. 2007 Sep 12;27(37):10000-6. doi: 10.1523/JNEUROSCI.2849-07.2007. PMID 17855614
- [Result] Harris RE, Sundgren PC, Craig AD, Kirshenbaum E, Sen A, Napadow V, Clauw DJ. Elevated insular glutamate in fibromyalgia is associated with experimental pain. Arthritis Rheum. 2009 Oct;60(10):3146-52. doi: 10.1002/art.24849. PMID 19790053
- [Result] Napadow V, LaCount L, Park K, As-Sanie S, Clauw DJ, Harris RE. Intrinsic brain connectivity in fibromyalgia is associated with chronic pain intensity. Arthritis Rheum. 2010 Aug;62(8):2545-55. doi: 10.1002/art.27497. PMID 20506181
- See also: Chronic Pain and Fatigue Research Center — http://www.med.umich.edu/painresearch/study/index.htm